CLINICAL TRIAL: NCT05746156
Title: Lymphatic Mapping for Image Guided Radiotherapy in Patients With Locally Advanced Cervical Cancer, a Feasibility Study
Brief Title: Lymphatic Mapping for Image Guided Radiotherapy in Patients With LACC - a Feasibility Study
Acronym: LaMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Dr Shandra Bipat PhD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL9323
Record Dates: First submitted 2023-02-17; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Locally Advanced Cervical Cancer

STUDY DESIGN:
Masking Description: Results of the lymphatic map will be blinded to the radiation oncologist
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lymphatic map (Experimental): Lymphatic mapping will be performed
  Interventions: Diagnostic Test: lymphatic mapping

INTERVENTIONS:
Diagnostic Test: lymphatic mapping — 1. Peritumoral injection of [99mTc]Tc-nanocolloid in 6-8 evenly distributed depots on both sides of the tumor, during investigation under anaesthesia. Number of depots depending on the size and localisation of the tumor.
  2. Planair and SPECT/CT imaging van de abdomen/pelvis 3h and 12-24h after injection at the department of radiology and nucleair medicine.

SUMMARY:
Lymphatic mapping is a procedure in which all lymph nodes with drainage from the primary tumor, i.e. all nodes with potential (micro)metastases, can be imaged. These nodes are not necessarily suspicious on other imaging techniques.

The goal of this feasibility study is to

1. investigate the feasibility of the lymphatic mapping procedure in locally advanced cervical cancer
2. study the agreement of the lymphatic map with the radiotherapy treatment plan including previous imaging (MRI / CT / FDG-PET/CT)

DETAILED DESCRIPTION:
Study population:

Aged ≥18 years, with locally advanced cervical cancer, that will be planned for radiotherapy.

Intervention (if applicable): Lymphatic mapping will be performed on all study patients during the standard investigation under anaesthesia, to ensure painless injection of the radiopharmaceutical. Patients will receive 6-8 depots of [99mTc]Tc-nanocolloid peritumoral. Planar and SPECT/CT gamma camera images will be made at the department of Radiology and Nuclear medicine 3 hours and 12-24 hours after administration of the radiopharmaceutical. All radioactive lymph nodes will be included in the lymphatic map.

The radiation oncologist will determine the radiation therapy treatment plan blinded to the data of the lymphatic mapping. The lymphatic map will be compared to the radiation treatment plan and previous imaging (MRI / CT / FDG-PET/CT).

Main study parameters/endpoints:

1. Is it feasible to perform lymphatic mapping in locally advanced cervical cancer? Is there visualisation of (multiple) lymph nodes in both sides of the tumor?
2. Are all visible lymph nodes (nodes at risk) included in the standard radiotherapy treatment plan?

ELIGIBILITY:
Inclusion Criteria:

Histologically proven locally advanced cervical cancer [FIGO stage IIB-IVA]. >18 years old. Treatment with curative (chemo)radiation. Signed informed consent.

Exclusion Criteria:

Pregnancy. Administration of the radioactive tracer cannot be ensured properly due to obesity Patients with tumors in which no circumferential injection of [99mTc]Tc-nanocolloid is possible due to the size or position of the tumor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Is it feasible to perform lymphatic mapping in locally advanced cervical cancer? Is there visualisation of (multiple) lymph nodes in both sides of the tumor? | 2 years
  feasibiliy

SECONDARY OUTCOMES:
Are all visible lymph nodes (nodes at risk) included in the standard radiotherapy treatment plan? | 2 years
  comparison to RT treatment plan

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC University of Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adam JA, Poel E, van Eck-Smit BLF, Mom CH, Stalpers LJA, Stoker J, Bipat S. Lymphatic mapping for image-guided radiotherapy in patients with locally advanced uterine cervical cancer: a feasibility study. EJNMMI Res. 2023 Jun 12;13(1):58. doi: 10.1186/s13550-023-00989-0. PMID 37306763